CLINICAL TRIAL: NCT07202286
Title: Comparing Physician and Artificial Intelligence Chatbot Responses to Frequently Asked Questions From Osteoarthritis Patients: a Prospective Cross-sectional Study
Brief Title: Comparing Physician and Artificial Intelligence Chatbot Responses to Frequently Asked Questions From Osteoarthritis Patients
Acronym: PARTICIPATE
Status: Completed | Type: Observational
Sponsor: Canisius-Wilhelmina Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 075-2023
Record Dates: First submitted 2025-09-30; First posted 2025-10-01 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Osteo Arthritis Knee and Hip; Artificial Intelligence (AI); Acceptability; Accuracy; Chatbot
Keywords: chatGPT; Osteoarthritis; Acceptability; Accuracy; Artificial Intelligence; Cross-sectional
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aimed to compare the patient acceptability (preference, length, and difficulty) and accuracy of Chat-Generative Pre-Trained Transformer (ChatGPT) responses to questions from people with osteoarthritis (OA) with physician responses.

DETAILED DESCRIPTION:
This was a cross-sectional study where participants were invited by e-mail to participate in the questionnaire to compare Chatbot responses to physician responses.

ELIGIBILITY:
Inclusion Criteria:

* all individuals visiting the Department of Orthopedics in the Canisius Wilhelmina Hospital, a district general hospital in Nijmegen, The Netherlands, diagnosed with knee or hip OA between March 2023 and March 2024

Exclusion Criteria:

* partly completion of the questionnaire

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: There were two groups of participants: 1) a panel of people with OA evaluating the preference, length, and difficulty, and 2) a panel of experts in the field of OA evaluating the accuracy of the responses
Sampling Method: Non-Probability Sample
Enrollment: 286 (Actual)
Dates: Start 2024-05-22 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-06-05 (Actual)

PRIMARY OUTCOMES:
Preferred response | From invitation until the end of the study at two weeks
  Binary outcome, chatbot or physician response. This was an average based on the preferences on the 7 FAQs.

SECONDARY OUTCOMES:
Rating of length | From invitation until the end of the study at two weeks
  Rating of both responses (chatbot and physician response) included 'too short', 'good', and 'too long'.
Rating of difficulty | From invitation until the end of the study at two weeks
  Rating of difficulty included 'too easy', 'good', and 'too difficult' for both responses.
Accuracy | From invitation until the end of the study at two weeks
  Accuracy of the responses included the options 'Completely incorrect,' 'partly incorrect, ' 'approximately equally correct and incorrect,' 'mostly correct,' 'completely correct'.

OTHER OUTCOMES:
Number of words of the responses | This was determined before the study started

CONTACTS AND LOCATIONS:
Locations (1):
- Canisius Wilhelmina Hospital, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
The dataset supporting the conclusions of this study is available from the corresponding author upon reasonable request.